CLINICAL TRIAL: NCT07074353
Title: A Randomized, Multicenter Clinical Study of Irinotecan Liposomes in Total Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Brief Title: Irinotecan Liposomes in Total Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Acronym: CinClare-2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, Coordinating Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CinClare-2
Record Dates: First submitted 2025-07-08; First posted 2025-07-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRI-TNT (Experimental): Irinotecan Liposomes+Long-course concurrent chemoradiotherapy followed by consolidation chemotherapy
  Interventions: Drug: NALIRI; Radiation: LCRT; Drug: FOLFOX
- TNT (Placebo Comparator): Long-course concurrent chemoradiotherapy followed by consolidation chemotherapy
  Interventions: Radiation: LCRT; Drug: FOLFOX

INTERVENTIONS:
Drug: NALIRI — Irinotecan liposomes
  Arms: NALIRI-TNT
Radiation: LCRT — Long-course concurrent chemoradiotherapy
Drug: FOLFOX — Fluorouracil/Leucovorin, Oxaliplatin (5-FU/LV, OX)

SUMMARY:
This study enrolled patients with locally advanced rectal cancer. The experimental group received irinotecan liposomes combined with standard total neoadjuvant therapy (TNT), while the control group received standard TNT. The study endpoints were the complete response rate (cCR + pCR), 3-year event-free survival (EFS) rate, and overall survival (OS). The aim was to compare the efficacy and safety of irinotecan liposomes combined with or without standard TNT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years, both male and female are eligible;
2. Histologically confirmed rectal adenocarcinoma;
3. Clinical stage assessed by MRI as T3-4 or N+ (according to the 8th edition of the AJCC);
4. Distance from the lower edge of the tumor to the anal verge ≤ 10 cm;
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1;
6. UGT1A1*6 and UGT1A1*28 gene phenotypes are either wild-type (GG+6/6) or single-site mutant (GG+6/7 or GA+6/6);
7. No prior anti-tumor treatment for rectal cancer, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.;
8. Normal function of major organs.

Exclusion Criteria:

1. Previous or ongoing treatment for rectal cancer, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.
2. Known MSI-H (high microsatellite instability) by genetic testing or dMMR (deficient mismatch repair) by immunohistochemistry.
3. Known hypersensitivity, allergic reaction, or contraindication to irinotecan liposomes/vehicle, irinotecan, other liposomal products, 5-FU, leucovorin, oxaliplatin, or any of these agents.
4. Uncontrolled cardiac symptoms or disease.
5. Severe infection (CTCAE > Grade 2) within 4 weeks prior to the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, or infectious complications; baseline chest imaging showing active pulmonary inflammation; signs and symptoms of infection within 14 days prior to the first use of the study drug or requiring oral or intravenous antibiotic therapy, excluding prophylactic use of antibiotics.
6. Severe gastrointestinal dysfunction (inflammation or diarrhea greater than Grade 1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response rate（CR） | cCR: before the surgery, and up to 4 weeks after the end of completation of total neoadjuvant therapy (TNT) for cCR. pCR: after the surgery.
  Clinical Complete Response rate（cCR）+ Pathological Complete Response rate （pCR）

SECONDARY OUTCOMES:
3-year event-free survival (3y-EFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No